CLINICAL TRIAL: NCT02272855
Title: A Phase II Study of Combination Treatment With HF10, a Replication-competent HSV-1 Oncolytic Virus, and Ipilimumab in Patients With Stage IIIB, Stage IIIC, or Stage IV Unresectable or Metastatic Malignant Melanoma
Brief Title: A Study of Combination Treatment With HF10 and Ipilimumab in Patients With Unresectable or Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takara Bio Inc. (Industry)
Collaborators: Theradex (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T14-10682
Record Dates: First submitted 2014-10-09; First posted 2014-10-23 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Malignant Melanoma
Keywords: HF10; HSV-1; Ipilimumab; Oncolytic virus; Phase II; Stage IIIB melanoma; Stage IIIC melanoma; Stage IV melanoma; Unresectable malignant melanoma; Metastatic malignant melanoma; Combination treatment; Intratumoral injection
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HF10 plus ipilimumab (Experimental)
  Interventions: Biological: HF10 plus Ipilimumab

INTERVENTIONS:
Biological: HF10 plus Ipilimumab — Patients will receive the dose of 1 x 10^7 TCID50/mL HF10 (for a total of 6 injections; the first 4 injections at 1-week intervals; the remaining 2 injections at 3-week intervals) and ipilimumab at 3 mg/kg ipilimumab (for a total of 4 intravenous infusions, each administered at 3-week intervals).
  Other Names: YERVOY (for ipilimumab)

SUMMARY:
The purpose of this study is to determine if HF10 in combination with ipilimumab is effective in patients with stages IIIB, IIIC, or IV unresectable or metastatic melanoma.

DETAILED DESCRIPTION:
The study is designed to assess efficacy and safety with repeated administration of intratumoral injections of HF10 at 1x10^7 TCID50/mL in combination with intravenous infusions of 3mg/kg ipilimumab. This is a single arm, open label Phase II trial, to evaluate the efficacy, safety and tolerability of HF10 treatment in combination with administration of the immunologic checkpoint inhibitor, ipilimumab (anti-CTLA-4 monoclonal antibody). The study population will include patients with Stage IIIB, IIIC or IV unresectable or metastatic malignant melanoma who are ipilimumab-eligible.

Patients will receive the dose of 1 x 10^7 TCID50/mL HF10 (for a total of 6 injections; the first 4 injections at 1-week intervals; the remaining 2 injections at 3-week intervals) + ipilimumab at 3 mg/kg ipilimumab (for a total of 4 intravenous infusions, each administered at 3-week intervals).

Following combination therapy, patients may continue to receive the same dose level of HF10 (1 x 10^7 TCID50/mL) alone for up to an additional 13 injections (total of 19 injections = 1 year) if they have tolerated the study treatment, are responding, have stable disease, or have progressive disease that is not clinically significant in the judgment of the Investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have Stage IIIB, IIIC or IV melanoma, which is unresectable/unresected or histologically confirmed diagnosis of metastatic malignant melanoma.
2. Patients must have measurable non-visceral lesion(s) that are evaluable by the modified World Health Organization (mWHO) criteria and immune-related response criteria (irRC).
3. Patients must be ≥ 18 years of age.
4. Patients must have a life expectancy ≥ 24 weeks.
5. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
6. Patients must have adequate hepatic function, defined as

   * Total bilirubin levels ≤ 1.5 x upper limit of normal [ULN] (except for patients with Gilbert's Syndrome, who must have a total bilirubin of less than 3.0 mg/dL)
   * AST/ALT levels ≤ 2.5 x ULN, or ≤ 5 x ULN if liver metastases are present.
7. Patients must have adequate renal function, defined as serum creatinine ≤ 1.5 x ULN or creatinine clearance (calculated) ≥ 60 mL/min/1.73 m2 for patients with creatinine > 1.5 x ULN.
8. Patients must have adequate bone marrow function, defined as

   * Absolute neutrophil count ≥1,500/µL and
   * Platelet count ≥ 75,000/ µL
9. Patients must have no known bleeding diathesis or coagulopathy that would make intratumoral injection or biopsy unsafe.
10. Patients must be ipilimumab-eligible. (This includes: 1) patients previously untreated with ipilimumab; 2) patients previously treated (more than 1 year previously) with ipilimumab using a route of administration other than intravenous infusion; and 3) patients previously treated with antitumor agents other than intravenous ipilimumab).
11. Men and women of childbearing potential must agree to use adequate contraception from the time of consent through 30 days after final study treatment.
12. Females of childbearing potential must have a negative urine or serum pregnancy test within one week prior to start of treatment.
13. Patients must be able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

1. Patients receiving chemotherapy or radiotherapy within 4 weeks of injection of HF10, or history of Grade 4 adverse events or presence of adverse events Grade 2 or greater, except alopecia, resulting from anticancer agents administered more than 4 weeks prior to HF10 injection.
2. Patients receiving anti-herpes medication within 1 week prior to initiating HF10 treatment.
3. Patients with a history of significant tumor bleeding, or coagulation or bleeding disorders.
4. Patients with target tumors that could potentially invade a major vascular structure (e.g., innominate artery, carotid artery), based on unequivocal imaging findings.
5. Patients with Grade 2 or greater pre-existing neurologic abnormalities (CTCAE version 4.0), including Grade 2 or greater peripheral neuropathy caused by previous treatments.
6. Patients with clinically evident Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), Hepatitis C virus (HCV), or Epstein-Barr virus (EBV) infection are excluded.
7. Medical history of autoimmune disease (e.g., Crohn's disease, ulcerative colitis) or other diseases requiring systemic glucocorticoid or immunosuppressive therapy.
8. Patients who were previously treated with ipilimumab administered by intravenous infusion.
9. Concurrent use of any other investigational agents.
10. Patients with active CNS metastases or carcinomatous meningitis, except patients with CNS lesions that have been treated and have no evidence of progression in the brain on CT/MRI for ≥ 3 months.
11. Pregnant or breastfeeding women; women desiring to become pregnant within the timeframe of the study are also excluded.
12. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-04-30 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Best overall response rate (BORR) | at 24 weeks

SECONDARY OUTCOMES:
Adverse Event Summaries, Vital Signs, and Laboratory Parameters as a Measure of Safety and Tolerability | until Week 24
  Adverse events will be evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE version 4.0).
Objective response rate (ORR) | at Weeks 12, 18, and 24
Progression-free survival (PFS) | for 1 year
Durable response rate (DRR) | for 1 year
1-year survival rate | at 1 year
Accumulation of Lymphocytes in the Tumor by using Core Biopsy Samples | pre-treatment screening and Week 24
Change in Cytokine Profiles by using Peripheral Blood Samples | pre-treatment screening and Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Robert Andtbacka, Principal Investigator — University of Utah
Locations (8):
- United States (8):
  - Clinical Site, San Francisco, California
  - Clinical Site, Atlanta, Georgia
  - Clinical Site, Portland, Oregon
  - Clinical Site, Bethlehem, Pennsylvania
  - Clinical Site, Hershey, Pennsylvania
  - Clinical Site, Dallas, Texas
  - Clinical Site, Houston, Texas
  - Clinical Site, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Watanabe D, Goshima F. Oncolytic Virotherapy by HSV. Adv Exp Med Biol. 2018;1045:63-84. doi: 10.1007/978-981-10-7230-7_4. PMID 29896663